CLINICAL TRIAL: NCT06823076
Title: Impact of the COVID-19 Pandemic on Central Precocious Puberty: a Retrospective Cohort Study from Turkey
Acronym: COVID-19-PP
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, gulcan seymen, MD, Umraniye Education and Research Hospital
Other Study IDs: 406240
Record Dates: First submitted 2025-02-11; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2023-02

CONDITIONS: COVID19- Infection with SARS-CoV-2 Virus
Keywords: Central precocious puberty, COVID-19 pandemic, GnRH analogs, pediatric endocrinology, lifestyle changes
MeSH Terms: conditions — Puberty, Precocious; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- prepandemic and pandemic precocious puberty groups were compared

SUMMARY:
Objective: This study investigates the clinical and demographic characteristics of girls diagnosed with central precocious puberty (CPP) in the pre-pandemic and pandemic periods to assess potential changes during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Methods: A retrospective cohort study was conducted on patients admitted to the Pediatric Endocrinology Departments of two centers in Turkey. Girls treated with GnRH analogs between March 2018 and 2022 were categorized into two groups: the pre-pandemic group (2018-2020) and the pandemic group (2020-2022). Clinical, anthropometric, and hormonal data were analyzed. Patients with organic lesions, genetic conditions, or medications affecting puberty were excluded.

ELIGIBILITY:
Inclusion Criteria (Who Can Participate?)

Girls: Tanner stage ≥2 before age 8 peak LH > on gnrh analog test, basal Lh >0,3

Patients with organic lesions (e.g., hypothalamo-pituitary tumors), congenital malformations, oncological diseases, neurosurgical or genetic disorders, or medications affecting puberty were excluded from the study

Max Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study included patients admitted to the Pediatric Endocrinology Departments of Umraniye Training and Research Hospital and Suleyman Demirel University, located in two different cities in Turkey. These patients were diagnosed with precocious puberty and treated with GnRH analogs before and after the COVID-19 pandemic. The patients were categorized into two groups: the pre-pandemic group (admitted and started GnRH analog treatment between March 2018 and March 2020) and the pandemic group (admitted and started GnRH analog treatment between March 2020 and March 2022), covering 24 months before and after the start of the pandemic lockdown
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Mean Age at Pubertal Onset | 4 years
  Mean Age at Pubertal Onset
  Description: The mean age at pubertal onset will be compared between pre-pandemic and post-pandemic periods in both girls and boys.
  Time Frame: At baseline. Method of Measurement: Tanner staging, LH/FSH levels, and bone age assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- the Pediatric Endocrinology Departments of Umraniye Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and institutional policies. Only aggregated study results will be published in peer-reviewed journals."